CLINICAL TRIAL: NCT02773459
Title: Phase Ib Study of MEK162 in Combination With Capecitabine in Gemcitabine-pretreated Advanced Biliary Tract Cancer
Brief Title: MEK162 in Combination With Capecitabine in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTC-MEK162
Record Dates: First submitted 2016-05-13; First posted 2016-05-16 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — binimetinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 part (Experimental): to assess the maximal tolerated dose (MTD) of MEK162+Capecitabine combination
  Interventions: Drug: MEK162+capecitabine
- Expansion part (Experimental): to assess the efficacy (PFS) of MEK162+Capecitabine combination
  Interventions: Drug: MEK162+capecitabine

INTERVENTIONS:
Drug: MEK162+capecitabine — In phase 1 part: capecitabine(mg/m2) will be given twice a day, 2 week on/1week off Q 3weeks + MEK162 twice a day, continuously, starting at 1000mg/m2 and 30mg/m2 respectively. Expansion part will be treated with the dose found at phase 1 part.
  Other Names: MEK162, xeloda

SUMMARY:
This study is to test the efficacy of MEK162 plus capecitabine in gemcitabine-pretreated advanced biliary tract cancer, and to explore the predictive biomarkers for future large-scale clinical trials using this combination.

DETAILED DESCRIPTION:
Biliary tract cancer is one of rare cancers, which is relatively more frequent in east Asia. The frequency of KRAS mutation and/or BRAF mutation is reported at 40 to 60%. The prognosis is still very poor, with only limited treatment options. The most commonly used 1st-line chemotherapy is gemcitabine+cisplatin combination. In gemcitabine-pretreated advanced biliary tract cancer, fluoropyrimidine-based chemotherapy is used. However, the overall survival with these cytotoxic chemotherapies is still only about 8-10 months, calling for urgent development of efficient treatment options.

Recently, mitogen-activated extracellular signal regulated kinase kinase (MEK) inhibition was shown to have antitumor effects in KRAS mutated biliary tract cancers in preclinical model. In phase II study of MEK inhibitor (selumetinib) in metastatic biliary tract cancers, selumetinib displayed interesting activity and acceptable tolerability.

MEK162 is an oral, highly selective MEK inhibitor. It was shown to promote apoptosis and in vivo antitumor activity against human biliary tract cancer cell lines. So far, there has been no study to test the MEK inhibitor mainly in gemcitabine-pretreated advanced biliary tract cancer, especially in combination of capecitabine chemotherapy.

The aim of this study is to test the efficacy of MEK162 plus capecitabine in gemcitabine-pretreated advanced biliary tract cancer, and to explore the predictive biomarkers for future large-scale clinical trials using this combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically / cytologically verified, non-resectable, recurrent, or metastatic biliary tract carcinoma including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma
* Patients who have previously treated with gemcitabine-based chemotherapy (Prior treatment regimen up to 2 is allowed)
* Patients must have measurable or evaluable disease by RECIST 1.1
* Eastern Eastern Cooperative Oncology Group (ECOG) performance status: 0, 1
* Age ≥ 20 years
* Adequate bone marrow function defined as: Hb ≥ 8 g/dl, absolute neutrophil count (ANC) ≥ 1500/microliter (mcL), Platelets ≥ 100 x10^3/mcL
* Adequate renal function defined as serum creatinine < 1.6 mg/dl and/or measured creatinine clearance from 24-hour urine collection of ≥ 60 ml/min
* Adequate hepatic function defined as total bilirubin ≤ 2 mg/dl, alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN)
* Patients with biliary obstruction can join if bilirubin corrects to required limit after adequate biliary drainage
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to study treatment
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of another active cancer that may influence patient outcome, except for nonmelanoma skin carcinoma, melanoma in-situ, in-situ carcinoma of the cervix curatively treated, treated superficial bladder cancer, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment prostate surface antigen (PSA) that is non-detectable
* Known brain metastases or primary central nervous system tumors with seizures that are not well controlled with standard medical therapy
* Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements
* Known HIV positive patient
* Significant cardiovascular disease including congestive heart failure (New York Heart Association Class II or higher) or active angina pectoris
* Uncontrolled diabetes mellitus
* History of a myocardial infarction within 6 months
* History of a stroke or transient ischemic attack within 6 months
* Clinically significant peripheral vascular disease
* Major surgical procedure within 4 weeks
* Uncontrolled infection
* Known or suspected allergy to capecitabine
* Pregnant (positive pregnancy test)
* Breast-feeding should be discontinued if a nursing mother is to be treated on clinical trial
* Any condition that impairs patient's ability to swallow whole pills
* Malabsorption problem that may limit or inhibit the absorption of MEK162
* History of any organ or bone marrow transplant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 6 months
  MTD in all treated population (Phase 1 part)
Progression-free survival (PFS) | 3 months
  PFS in all treated population (Expansion part)

SECONDARY OUTCOMES:
Dose-limiting Toxicity (DLT) | 6 months
  DLT in all treated population, according to NCI-CTCAE v 4.0 (Phase 1 part)
Recommended Phase 2 Dose (RP2D) | 6 months
  RP2D to be used at Expansion part (Phase 1 part)
Response rate | 6 months
  Response rate in all treated patients (Expansion part)
Overall survival (OS) | 1 year
  OS in all treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JW, Lee KH, Kim JW, Suh KJ, Nam AR, Bang JH, Bang YJ, Oh DY. Enhanced antitumor effect of binimetinib in combination with capecitabine for biliary tract cancer patients with mutations in the RAS/RAF/MEK/ERK pathway: phase Ib study. Br J Cancer. 2019 Aug;121(4):332-339. doi: 10.1038/s41416-019-0523-5. Epub 2019 Jul 17. PMID 31312030